CLINICAL TRIAL: NCT02250807
Title: A Phase 3, Multicenter, Open-Label, Single-Arm Study to Investigate the Efficacy and Safety of a 12-Week Regimen of Simeprevir in Combination With Sofosbuvir in Treatment-Naive or -Experienced Subjects With Chronic Genotype 4 Hepatitis C Virus Infection
Brief Title: Efficacy and Safety Study of Simeprevir in Combination With Sofosbuvir in Subjects With Chronic Genotype 4 Hepatitis C Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR105429; TMC435HPC3021 (Other: Janssen R&D Ireland); 2014-003446-27 (EudraCT Number); NCT02256176 (obsolete NCT alias)
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Hepatitis C; Genotype 4 Chronic Hepatitis C
Keywords: Chronic hepatitis C; Genotype 4 chronic hepatitis C; Simeprevir; Sofosbuvir
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Simeprevir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simeprevir and Sofosbuvir (Experimental): Subjects will receive oral capsule of Simeprevir 150 milligram (mg) along with oral tablet of sofosbuvir 400 mg, once a day from Day 1 up to Week 12.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Simeprevir — Subjects will receive oral capsule of Simeprevir 150 mg, once a day from Day 1 up to Week 12.
  Other Names: TMC435
Drug: Sofosbuvir — Subjects will receive oral tablet of sofosbuvir 400 mg, once a day from Day 1 up to Week 12.

SUMMARY:
The purpose of this study is to show superiority of simeprevir (SMV) in combination with sofosbuvir for 12 weeks versus a historical control. Historical control will be a composite of the observed historical sustained virological response at Week 12 (SVR12) rates of SMV in combination with (pegylated) interferon (PegIFN)/ribavirin (RBV) of the subpopulations in study HPC3011 (NCT01567735) and will depend on the percentage of treatment-naive, prior relapser, prior non-responder, interferon (IFN)-intolerant and other subjects enrolled in this study.

DETAILED DESCRIPTION:
This is a Phase 3, open-label (all people know the identity of the intervention), single-arm, multicenter study (conducted at multiple sites). The study consists of 3 periods: a Screening period (up to 4 weeks), Treatment period (12 Weeks) and Post treatment follow-up period (until 24 weeks after end of treatment). The duration of the subjects' participation will be approximately 40 weeks. In the treatment period subjects will receive oral capsule simeprevir along with oral tablet sofosbuvir once daily for 12 weeks. Primarily efficacy will be evaluated as percentage of subjects with sustained virologic response at Week 12 after the end of treatment. Subjects' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with confirmed hepatitis C virus (HCV) with HCV RNA greater than (>) 10000 international unit per milliliter (IU/mL)
* Subjects who are treatment naive or treatment-experienced.
* Subjects must have documentation of a liver biopsy or fibroscan or agree to have one during screening
* Subjects with cirrhosis must have an hepatic imaging procedure (ultrasound, CT scan or magnetic resonance imaging [MRI]) within 6 months before the screening visit (or during the screening period) with no findings suspicious for hepatocellular carcinoma (HCC)
* Women of childbearing potential or men with a female partner of childbearing potential must agree to use an effective form of contraception, or not be heterosexually active, or of nonchildbearing potential

Exclusion Criteria:

* Evidence of clinical hepatic decompensation
* Any liver disease of non-HCV etiology
* Subjects with a past history of treatment with an approved or investigational DAA
* Co-infection with human immunodeficiency virus (HIV) type 1 or type 2 (HIV-1 or HIV-2) (positive HIV-1 or HIV-2 antibodies test at screening)
* Infection/co-infection with HCV non-genotype 4

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trials, Study Director — Janssen R&D Ireland
Locations (6):
- Spain (6):
  - Badalona
  - Barcelona
  - Madrid
  - Santander
  - Seville
  - Valencia

REFERENCES:
- [Derived] Buti M, Calleja JL, Lens S, Diago M, Ortega E, Crespo J, Planas R, Romero-Gomez M, Rodriguez FG, Pascasio JM, Fevery B, Kurland D, Corbett C, Kalmeijer R, Jessner W. Simeprevir in combination with sofosbuvir in treatment-naive and -experienced patients with hepatitis C virus genotype 4 infection: a Phase III, open-label, single-arm study (PLUTO). Aliment Pharmacol Ther. 2017 Feb;45(3):468-475. doi: 10.1111/apt.13883. Epub 2016 Nov 29. PMID 27896822

RESULTS

PARTICIPANT FLOW:
Groups:
- SMV+SOF 12 Weeks: Participants received oral capsule of simeprevir (SMV) 150 milligram (mg) and an oral tablet of sofosbuvir (SOF) 400 mg, once a day from Day 1 through Week 12.
Period: Overall Study
Arm/Group | SMV+SOF 12 Weeks
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SMV+SOF 12 Weeks
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 51 [29 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After End of Treatment (EOT) (SVR12)
Description: SVR12 is defined as the percentage of participants with hepatitis C virus ribonucleic acid (HCV RNA) less than (<) lower limit of quantification (LLOQ; 15 international unit per milliliter [IU/mL]) detectable or undetectable 12 weeks after actual EOT.
Time Frame: 12 weeks after EOT
Population: Intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study medication (SMV and/or SOF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SMV+SOF 12 Weeks
Number analyzed (Participants) | 40
percentage of participants | 100 [91.2 to 100]

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After End of Therapy (SVR4)
Description: SVR4 is defined as the percentage of participants with hepatitis C virus ribonucleic acid (HCV RNA) less than (<) lower limit of quantification (LLOQ; 15 international unit per milliliter [IU/mL]) detectable or undetectable 4 weeks after actual EOT.
Time Frame: 4 weeks after EOT
Population: ITT population included all randomized participants who received at least 1 dose of study medication (SMV and/or SOF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SMV+SOF 12 Weeks
Number analyzed (Participants) | 40
percentage of participants | 100 [91.2 to 100]

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After End of Therapy (SVR24)
Description: Participants were considered to have reached SVR24, if at the time point of SVR24 (that is [i.e.], 24 weeks after the end of treatment [EOT]) the following condition has been met: HCV RNA < lower limit of quantification (LLOQ), i.e., 15 IU/mL, detectable or undetectable.
Time Frame: At 24 weeks after EOT
Population: ITT population included all randomized participants who received at least 1 dose of study medication (SMV and/or SOF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SMV+SOF 12 Weeks
Number analyzed (Participants) | 40
percentage of participants | 100 [91.2 to 100.0]

4. Secondary Outcome: Percentage of Participants With On-treatment Virologic Response of Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
Description: Percentage of participants with HCV RNA less than (<) 15 IU/mL undetectable or detectable or detectable /undetectable at specific time points were observed.
Time Frame: Week 2, 3, 4, 12 and EOT
Population: ITT population included all randomized participants who received at least 1 dose of study medication (SMV and/or SOF).
Measure: Number; unit: percentage of participants
Arm/Group | SMV+SOF 12 Weeks
Number analyzed (Participants) | 40
percentage of participants
  Week 2: < 100 IU/mL | 87.5
  Week 2: < 15 IU/mL undetectable/detectable | 40.0
  Week 2: < 15 IU/mL undetectable | 17.5
  Week 3: < 100 IU/mL | 100.0
  Week 3: < 15 IU/mL undetectable/detectable | 82.5
  Week 3: < 15 IU/mL undetectable | 40.0
  Week 4: < 100 IU/mL | 100.0
  Week 4: < 15 IU/mL undetectable/detectable | 87.5
  Week 4: < 15 IU/mL undetectable (RVR) | 65.0
  Week 12: < 100 IU/mL | 100.0
  Week 12: < 15 IU/mL undetectable/detectable | 100.0
  Week 12: < 15 IU/mL undetectable | 100.0
  End of Treatment (EOT): < 100 IU/mL | 100.0
  EOT: < 15 IU/mL undetectable/detectable | 100.0
  EOT: < 15 IU/mL undetectable | 100.0

5. Secondary Outcome: Percentage of Participants With On-Treatment Failure
Description: Participants were considered on-treatment failures if they have at EOT (confirmed) detectable HCV RNA, i.e., <LLOQ detectable or >=LLOQ.
Time Frame: through 12 weeks (EOT)
Population: ITT population included all randomized participants who received at least 1 dose of study medication (SMV and/or SOF).
Measure: Number; unit: percentage of participants
Arm/Group | SMV+SOF 12 Weeks
Number analyzed (Participants) | 40
percentage of participants | 0

6. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: Participants with confirmed >1.0 log10 increase in HCV RNA from nadir or confirmed HCV RNA >100 IU/mL in participants who had previously achieved HCV RNA <LLOQ.
Time Frame: Up to follow-up Week 24
Population: ITT population included all randomized participants who received at least 1 dose of study medication (SMV and/or SOF).
Measure: Number; unit: percentage of participants
Arm/Group | SMV+SOF 12 Weeks
Number analyzed (Participants) | 40
percentage of participants | 0

7. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Participants were considered to have viral relapse if they did not achieve SVR12 and meet the following conditions: 1) at EOT, HCV RNA less than (<)LLOQ, undetectable, and 2) during the follow-up period, HCV RNA greater than or equal to (>=)LLOQ.
Time Frame: Up to follow-up week 24
Population: ITT population included all randomized participants who received at least 1 dose of study medication (SMV and/or SOF).
Measure: Number; unit: percentage of participants
Arm/Group | SMV+SOF 12 Weeks
Number analyzed (Participants) | 40
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Up to EOT (Week 12)
Arm/Group | SMV+SOF 12 Weeks
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 17/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SMV+SOF 12 Weeks (N=40)
Headache (Nervous system disorders) | 8
Erythema (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Asthenia (General disorders) | 3
Catarrh (Respiratory, thoracic and mediastinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.